CLINICAL TRIAL: NCT04005235
Title: Assessment of Hemi-diaphragm Dysfunction After Upper Extremity Nerve Blocks Using Passive Oscillometry to Measure Lung Mechanics - A Pilot Study.
Brief Title: FOT Assessment of Hemi-diaphragm Dysfunction After Upper Extremity Nerve Blocks
Status: Terminated | Type: Observational
Why Stopped: Covid-19 pandemic, aerosol generating procedures
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Andrew Milne, Principal investigator, Nova Scotia Health Authority
Other Study IDs: FOTHDD1
Record Dates: First submitted 2019-06-17; First posted 2019-07-02 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Diaphragm Elevated; Paresis
Keywords: phrenic nerve; nerve block; ultrasonography; breath tests; oscillometry; brachial plexus
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Thorasys Tremoflo C-100 Airwave Oscillometry System (FOT) — Ultrasonography will be used to confirm hemidiaphragm dysfunction after brachial plexus nerve block. In subjects with U/S confirmed hemidiaphragm dysfunction, FOT measurements will be taken before and after nerve block and post-operatively after upper extremity surgery.
  Other Names: Hemidiaphragm ultrasonography

SUMMARY:
Upper extremity nerve blocks of the brachial plexus using local anesthetic can inadvertently affect the ipsilateral phrenic nerve and result in hemidiaphragm dysfunction. Ultrasonography is often used to assess for hemidiaphragm dysfunction after brachial plexus nerve blocks. Alternately, post-operative chest x-rays can also be used to document unilateral hemidiaphragm elevation secondary to phrenic nerve dysfunction. Newly developed passive breathing testing devices (Forced Oscillometry Technique - FOT) use small composite pressure waveforms (5-37Hz) imposed on top of normal breathing and measure the resulting reflected oscillations to assess the mechanical properties of the lungs. The lung resistance R(f) and reactance X(f) are automatically mathematically derived from the reflected pressure waveforms returning from the respiratory system to the FOT device. In this study, we will assess if FOT can be used to detect changes in lung mechanics (lung resistance R(f) and reactance X(f)) after ultrasound proven hemidiaphragm dysfunction secondary to brachial plexus nerve block.

DETAILED DESCRIPTION:
This study will be a prospective single centre observational trial using the Tremoflo Forced Oscillometry Technique (FOT) device to assess the changes in lung mechanical parameters after a brachial plexus nerve block with ultrasound confirmed hemidiaphragm dysfunction (HDD). The serial cohort in this study will be patients presenting for unilateral upper extremity surgery who are having a regional nerve block for anesthesia as part of their normal standard of care for surgery.

FOT has proven useful in monitoring and diagnosing small airway diseases such as asthma and chronic obstructive pulmonary disease, with further applications of FOT being researched in perioperative care applications including inhaled anesthesia and mechanical ventilation. The Tremoflo is useful in perioperative applications because it does not require active breathing maneuvers, unlike traditional pulmonary function tests like spirometry. This technique uses a composite waveform of (5,11,13,17,19,23, 29, 31 and 37 Hz) to measures respiratory system resistance (R(f), cmH2O/L/sec) as a function of frequency, reactance (X(f), cmH2O/L/sec) as a function of frequency, and the resonance frequency. Resistance increases as the airways narrow while a decrease in reactance represents stiffening or loss of inertia in the lungs. Resonance frequency is the frequency at which reactance as a function of frequency is equal to zero, it represents both the overall stiffening of the lungs and obstruction of the small airways. Oscillation, specifically at low frequencies (5-20Hz), measures the mechanical properties of the peripheral airways while oscillation at higher frequencies (>20Hz) measures the mechanical properties of the central and upper respiratory system, giving one a more complete overview of lung function.

Prior to study enrollment, patients will be screened and consented accordance to the department standard operating procedures. Demographic data will be collected including age, sex, weight, height, comorbid conditions to rule out any exclusion criteria.

A baseline ultrasonographic diaphragmatic assessment and Tremoflo measurement will be completed by all participants prior to nerve block. Any significant neurologic dysfunction, inability to visualize the diaphragm during sonographic assessment, pre-existing HDD or inability to use the Tremoflo device will result in withdrawing the patient from the study. Study participants will then receive a pre-operative ultrasound guided interscalene (ISB) or supraclavicular (SCB) brachial plexus block as per standard of care. A standard clinical mixture of ropivacaine and lidocaine will be injected incrementally at the discretion of the attending anesthesiologist.

An ultrasound machine with a linear transducer will be used to assess for hemidiaphragm dysfunction every 5 minutes after nerve block or until 30 minutes has elapsed. All subjects will lie in a semi-recumbent position. With the ultrasound set in B-mode, a longitudinal scan will be performed. The ABCDE (airway, breathing, circulation, disability and exposure) evaluation approach will be used which involves first placing the ultrasound probe along the anterior axillary line just below the 4th intercostal space on the ipsilateral side to the brachial plexus block. The movement of the pleura on top of the diaphragm will be visualized between the two ribs during normal breathing. The probe will then be moved caudally along the anterior axillary line to identify diaphragmatic thickening, where it will no longer be hidden under the pleura during inspiration, for examination. The diaphragm can then be easily distinguished from the adjacent intercostal muscles with visualization of the pleura just superficial to the diaphragm. The operator will visually examine the diaphragmatic muscle for the presence of a change in thickness. The probe will then be moved caudally, and when diaphragmatic thickening is clearly visualized in the zone of apposition, the thickness of diaphragm during expiration and deep inspiration will be determined using on-screen measurement caliper software built into ultrasound machine. Diaphragmatic dysfunction will be determined by intercostal diaphragm thickening based on validated criteria, with diaphragm thickening of less than 20% defined as dysfunction. The ultrasound image will be saved anonymously using a predefined study number.

The Tremoflo FOT assessment will be repeated after confirmed HDD by ultrasound criteria. All measurements will be taken while patients are in the semi-recumbent position, with the nostrils occluded using a disposable plastic clip that is routinely used with the Tremoflo device. A research team member will hold the Tremoflo device in the patients mouth and research staff or a Block room team member will gently support cheeks during all Tremoflo measurements. The research team will need to hold the device and support the cheeks as the patient will lack motor and sensory function due to the ISB/SCB nerve block.

After completion of the surgery, ultrasound diaphragmatic motion assessment and Tremoflo FOT measurement will be repeated in the post-operative care unit in the semi-recumbent position.

Subjective self-reported dyspnea (using the Modified Borg Dyspnea Scale, ordinal 0-10 scale with 0 = no breathlessness and 10 = maximal breathlessness) will be measured at baseline, then every 5 minutes after the nerve block until patient leaves for operating room or 30 minutes (whatever is earlier) and in the post-operative care unit at the time of ultrasound and FOT measurement.

The patients' data including age, sex, height (cm), weight (kg), body mass index (BMI) kg/m2, pertinent cardio-thoracic and neurologic medical history, nerve block details, ultrasound images and relevant anesthesia/surgical details (duration of surgical procedure, anesthetic type - regional anesthesia only vs. general anesthesia combined with upper extremity nerve block, muscle relaxant/reversal use - drug type and dose, airway management - oxygen face mask vs. laryngeal mask airway vs. tracheal tube) will be recorded for study purposes.

The co-primary outcome measures of this pilot study will be to determine:

1. Changes in FOT measured lung resistance R(f) after ultrasound confirmed HDD.
2. Changes in FOT measured lung reactance X(f) after ultrasound confirmed HDD.

The secondary outcomes will be to determine the incidence of subjective shortness of breath associated with an ISB/SCB and to determine FOT measured lung reactance and resistance changes after both a regional block and general anesthetic.

The sample size for the primary outcome measure was estimated using data from a study of FOT lung resistance changes at 5 Hz (R5) before and after patients underwent surgery for >2hrs under general anesthetic. Based on those outcomes, using a 1-sided T-test with alpha = 0.05, and beta = 0.8, sigma = 0.82, u1 = 2.31 and u2 = 2.75 the sample size required is 22 subjects. In order to account for drop-outs/attrition, 25 patients who experience HDD will be recruited to complete the study. The rate of HDD is different for the two standard types of upper extremity of nerve blocks used in this study. In the literature, ISB causes HDD in 100% of cases, while SCB incidence of HDD has been estimated at 50-67%. Historically, SCB are performed at a 4:1 ratio compared to ISB at our institution during normal surgical case loads. Based on these approximations, we anticipate recruiting 5 ISB (with 100% HDD) and 40 SCB (with a conservative estimated rate of 50% HDD) nerve block patients to meet our event rate based recruitment of a total of 25 patients who develop HDD for a total of 45 patients recruited.

Continuous respiratory variables automatically calculated by the Tremflo FOT device, such as respiratory system resistance, reactance, resonance frequency, tidal volume and respiratory rate will be expressed as mean and standard deviation or median and interquartile range dependant on their distribution. Changes in respiratory system resistance, reactance, resonance frequency, tidal volume and respiratory rate from before and after nerve block will be compared using ANOVA or appropriate non-parametric testing.

Participants will not be receiving any compensation, financial or otherwise, for their participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 y
* American Society of Anesthesiologists physical status class 1-3
* Undergoing upper extremity surgery which requires a pre-operative brachial plexus nerve block as part of their routine standard of care.

Exclusion Criteria:

* Contraindication to nerve block
* Pregnant patients
* Patient refusal or inability to provide informed consent
* Pre-existing hemidiaphragm dysfunction
* Any significant neurologic dysfunction, or inability to visualize the diaphragm during baseline sonographic assessment
* Inability to comply with FOT measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients requiring interscalene or supraclavicular nerve blocks as part of their routine standard of care, who develop ultrasound confirmed ipsilateral hemdiaphragm dysfunction.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Lung resistance - R(f) changes after brachial plexus block and ultrasound confirmed hemidiaphragm dysfunction | Baseline FOT measurements taken before nerve block and repeated immediately after ultrasound confirmation of hemidiaphragm dysfunction secondary to nerve block (onset of HDD estimated to be 5-30 mins after nerve block, per serial ultrasound assessments)
  Change from baseline FOT measured lung resistance R(f) in cmH2O/L/s
Lung reactance - X(f) changes after brachial plexus block and ultrasound confirmed hemidiaphragm dysfunction | Baseline FOT measurements taken before nerve block and repeated immediately after ultrasound confirmation of hemidiaphragm dysfunction secondary to nerve block (onset of HDD estimated to be 5-30 mins after nerve block, per serial ultrasound assessments)
  Change from baseline FOT measured lung reactance X(f) in cmH2O/L/s

SECONDARY OUTCOMES:
Subjective patient self reported dyspnea after brachial plexus nerve block | Every 5 minutes up to 30 minutes after the brachial plexus nerve block
  Using standard MBDS scale ("Modified Borg Dyspnea Scale", ordinal scale 0-10, 0 = no difficulty at all, 10 = maximal breathing difficulty)

OTHER OUTCOMES:
Post-operative Lung resistance - R(f) changes after brachial plexus block with ultrasound confirmed HDD and general anesthetic | In recovery room 30-60 mins after extubation, when alert enough to be compliant with testing.
  Change in FOT measured lung resistance R(f) after general anesthetic (cmH2O/L/s)
Post-operative Lung reactance - X(f) changes after brachial plexus block with ultrasound confirmed HDD and general anesthetic | In recovery room 30-60 mins after extubation, when alert enough to be compliant with testing.
  Change in FOT measured lung reactance X(f) after general anesthetic (cmH2O/L/s)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Mine, Principal Investigator — Staff
Locations (1):
- NSHA NHI site, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khurana J, Gartner SC, Naik L, Tsui BCH. Ultrasound Identification of Diaphragm by Novices Using ABCDE Technique. Reg Anesth Pain Med. 2018 Feb;43(2):161-165. doi: 10.1097/AAP.0000000000000718. PMID 29315130
- [Background] Gerscovich EO, Cronan M, McGahan JP, Jain K, Jones CD, McDonald C. Ultrasonographic evaluation of diaphragmatic motion. J Ultrasound Med. 2001 Jun;20(6):597-604. doi: 10.7863/jum.2001.20.6.597. PMID 11400933
- [Background] Kuzukawa Y, Nakahira J, Sawai T, Minami T. A Perioperative Evaluation of Respiratory Mechanics Using the Forced Oscillation Technique. Anesth Analg. 2015 Nov;121(5):1202-6. doi: 10.1213/ANE.0000000000000720. PMID 25839180
- [Background] Urmey WF, Talts KH, Sharrock NE. One hundred percent incidence of hemidiaphragmatic paresis associated with interscalene brachial plexus anesthesia as diagnosed by ultrasonography. Anesth Analg. 1991 Apr;72(4):498-503. doi: 10.1213/00000539-199104000-00014. PMID 2006740
- [Background] Knoblanche GE. The incidence and aetiology of phrenic nerve blockade associated with supraclavicular brachial plexus block. Anaesth Intensive Care. 1979 Nov;7(4):346-9. doi: 10.1177/0310057X7900700406. PMID 525758
- [Background] Neal JM, Moore JM, Kopacz DJ, Liu SS, Kramer DJ, Plorde JJ. Quantitative analysis of respiratory, motor, and sensory function after supraclavicular block. Anesth Analg. 1998 Jun;86(6):1239-44. doi: 10.1097/00000539-199806000-00020. PMID 9620512
- [Background] Mak PH, Irwin MG, Ooi CG, Chow BF. Incidence of diaphragmatic paralysis following supraclavicular brachial plexus block and its effect on pulmonary function. Anaesthesia. 2001 Apr;56(4):352-6. doi: 10.1046/j.1365-2044.2001.01708-2.x. PMID 11284823
- [Background] Oostveen E, MacLeod D, Lorino H, Farre R, Hantos Z, Desager K, Marchal F; ERS Task Force on Respiratory Impedance Measurements. The forced oscillation technique in clinical practice: methodology, recommendations and future developments. Eur Respir J. 2003 Dec;22(6):1026-41. doi: 10.1183/09031936.03.00089403. PMID 14680096
- [Background] Kanda S, Fujimoto K, Komatsu Y, Yasuo M, Hanaoka M, Kubo K. Evaluation of respiratory impedance in asthma and COPD by an impulse oscillation system. Intern Med. 2010;49(1):23-30. doi: 10.2169/internalmedicine.49.2191. Epub 2010 Jan 1. PMID 20045997